CLINICAL TRIAL: NCT02812186
Title: Effect of Deep Versus Moderate Neuromuscular Blockade on Peak Airway Pressures During Elective Laparoscopic Surgery
Brief Title: Deep Versus Moderate Neuromuscular Blockade During Laparoscopic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Ruchir Gupta, Clinical Assistant Professor, Stony Brook University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 823925
Record Dates: First submitted 2016-06-06; First posted 2016-06-24 (Estimated); Results first posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-03

CONDITIONS: Cholecystitis; Endometriosis; Bowel Obstruction; Fibroids; Prostate Cancer; Chronic Kidney Disease; Uterine Prolapse
Keywords: Neuromuscular blockade
MeSH Terms: conditions — Cholecystitis; Endometriosis; Intestinal Obstruction; Leiomyoma; Prostatic Neoplasms; Renal Insufficiency, Chronic; Uterine Prolapse | interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deep to Moderate NMB (Other): This group will undergo deep neuromuscular blockade, defined as post tetanic count (PTC) of 1 to 2, in the beginning portion of the surgery followed by a period of moderate blockade.
  Interventions: Procedure: Deep to Moderate NMB; Drug: Rocuronium
- Moderate to Deep NMB (Other): This group will undergo moderate neuromuscular blockade, defined as 1-2 twitches, in the beginning portion of the surgery followed by a period of deep blockade.
  Interventions: Procedure: Moderate to Deep NMB; Drug: Rocuronium

INTERVENTIONS:
Procedure: Deep to Moderate NMB — Rocuronium infusion will be paused and the Train of Four (TOF) monitor will be set to every 1-2 min. Once the patient has achieved a "moderate" NMB state (one to two twitches), the infusion of the muscle relaxant will be resumed at a low dose to maintain the patient at this level of blockade.
  Arms: Deep to Moderate NMB
Procedure: Moderate to Deep NMB — Rocuronium infusion will be increased in increments of 0.1-0.2 mg/kg/hr. and the TOF monitor will be set to every 1-2 min. Once the patient has no twitches and a PTC of 0-1 ("deep" NMB) the infusion will be adjusted to maintain the patient at this level of NMB.
  Arms: Moderate to Deep NMB
Drug: Rocuronium

SUMMARY:
This is a two period cross-over study randomizing patients undergoing laparoscopic surgery into 2 different groups: group 1 in which patients receive "deep neuromuscular blockade" in the beginning portion of their laparoscopic surgery followed by a period of "moderate blockade" and, group 2 in which patients receive "moderate neuromuscular blockade" in the beginning portion of their laparoscopic surgery followed by a period of "deep blockade". The deep neuromuscular block is defined as post tetanic count of 1 to 2 and the moderate neuromuscular block is defined as 1-2 twitches. In all patients, sugammadex is used to reverse the block at the end of surgery in order to obtain optimal extubating conditions.

DETAILED DESCRIPTION:
Neuromuscular blockade (NMB) is frequently utilized in laparoscopic procedures to improve surgical conditions by relaxing the abdominal muscles and thus facilitating insufflation with carbon dioxide to optimize surgical view. Increased airway pressures can lead to an increase in alveolar and perivascular edema, a decline in dynamic lung compliance and hypoxemia.

Several studies have investigated surgical view under deep vs. moderate neuromuscular blockade. Literature supports deep neuromuscular blockade providing better operating conditions/view by a surgeon and low airway pressures but, potentially, longer duration to extubation and worse respiratory mechanics at the end of anesthesia versus moderate neuromuscular blockade which shows worse operating conditions/view by a surgeon and worse airway pressures but possibly shorter duration to extubation and better respiratory mechanics at the end of anesthesia.

Thus, there is clearly equipoise with regard to the comparative effectiveness of deep vs medium NMB. Therefore, this study is designed to ascertain if a deep neuromuscular block will decrease the airway pressures in patients undergoing laparoscopic procedures compared to those under a moderate block. A reduction in airway pressures may lead to a decrease in the complications associated with elevated airway pressures including hypoxemia, total static lung compliance, alveolar edema, and long term morbidity. Additionally, the study aims to determine if time from administration of sugammadex to reversal is different between patients that have a moderate NMB as compared to a deep NMB.

ELIGIBILITY:
Inclusion Criteria:

* Each participant must be willing and able to provide written informed consent for the study.
* Each participant must be American Society of Anesthesiologists (ASA) class I, II or III.
* Each participant must be scheduled for elective laparoscopic surgery (this includes robotic laparoscopic surgery).
* Expected surgical duration of 60 min or longer

Exclusion Criteria:

* Inability to give informed oral or written consent
* Known or suspected neuromuscular disorders impairing neuromuscular function;
* True allergies as defined as hypotension, bronchospasm, or anaphylaxis to muscle relaxants, anesthetics or opioids
* A history (patient or family) of malignant hyperthermia
* A contraindication for neostigmine administration
* Renal insufficiency, as defined by serum creatinine levels at 2.5 fold the normal level
* Body mass index >40 kg/m^2
* Significant respiratory disease.
* Planned postoperative mechanical ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-12-27 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruchir Gupta, MD, Principal Investigator — Stony Brook Medicine
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No
Fully analyzed results may be shared with Merck Investigator Studies Program personnel after the study has completed

RESULTS

PARTICIPANT FLOW:
Groups:
- Deep to Moderate Neuromuscular Block (NMB): This group will undergo deep neuromuscular blockade, defined as post tetanic count (PTC) of 1 to 2, in the beginning portion of the surgery followed by a period of moderate blockade.
  Rocuronium
- Moderate to Deep NMB: This group will undergo moderate neuromuscular blockade, defined as 1-2 twitches, in the beginning portion of the surgery followed by a period of deep blockade.
  Rocuronium
Period: Period 1
Arm/Group | Deep to Moderate Neuromuscular Block (NMB) | Moderate to Deep NMB
Started | 40 | 39
Completed | 29 | 24
Not Completed | 11 | 15
Not completed — Post randomization screen failure | 5 | 9
Not completed — nonevaluable data sets | 6 | 6
Period: Period 2
Arm/Group | Deep to Moderate Neuromuscular Block (NMB) | Moderate to Deep NMB
Started | 29 | 24
Completed | 29 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deep to Moderate NMB | Moderate to Deep NMB | Total
Number analyzed (Participants) | 29 | 24 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (14.9) | 50.8 (15.4) | 51.8 (15.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 12 | 10 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 29 | 24 | 53
Procedure [Count of Participants; unit: Participants] — Surgical Procedure
  Participants
    General | 26 | 15 | 41
    General/Gynecology | 1 | 2 | 3
    Gynecology | 2 | 5 | 7
    Urology | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Peak Airway Pressures
Description: To determine if a deep NMB can lead to lower peak airway pressures in patients undergoing laparoscopic procedures when compared to a moderate NMB
Time Frame: Intra-operative, from intubation time to extubation time
Measure: Median (Inter-Quartile Range); unit: cm H2O
Groups:
- Deep NMB: This group underwent deep neuromuscular blockade, defined as post tetanic count (PTC) of 1 to 2, in the beginning portion of the surgery or during the second portion of the surgery
- Moderate NMB: This group underwent moderate neuromuscular blockade, defined as 1-2 twitches, in the beginning portion of the surgery or during the second period of the surgery
Arm/Group | Deep NMB | Moderate NMB
Number analyzed (Participants) | 53 | 53
cm H2O
  Mean | 25.5 [23.6 to 30.3] | 28.3 [23.9 to 35.0]
  Maximum | 28 [24 to 32] | 30 [27 to 36]
Statistical Analysis 1: Comparison: Deep NMB vs Moderate NMB; Test type: Superiority; p = 0.01, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Abdominal Insufflation Pressure
Description: To compare surgical operating condition by Abdominal Insufflation Pressure in patients undergoing laparoscopic procedures using deep NMB versus moderate NMB
Time Frame: Intra-operative, from intubation time to extubation time
Measure: Median (Inter-Quartile Range); unit: mmHg
Groups:
- Deep NMB: This group underwent deep neuromuscular blockade, defined as post tetanic count (PTC) of 1 to 2, in the beginning portion or during the second portion of the surgery
- Moderate NMB: This group underwent moderate neuromuscular blockade, defined as 1-2 twitches, in the beginning portion of the surgery or during the second portion of the surgery
Arm/Group | Deep NMB | Moderate NMB
Number analyzed (Participants) | 53 | 53
mmHg | 15 [14.8 to 15.2] | 15 [14.6 to 15.2]
Statistical Analysis 1: Comparison: Deep NMB vs Moderate NMB; Test type: Superiority; p = 0.28, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Surgical Rating Scale
Description: To compare surgical operating condition by Surgical Rating Scale (SRS) in patients undergoing laparoscopic procedures using deep NMB versus moderate NMB
  Surgical Rating Score scores are on a 1-5 scale with 1 = extremely poor conditions, 2 = poor conditions, 3 = adequate conditions, 4 = good conditions, 5= excellent conditions. Higher scores mean a better outcome.
Time Frame: Intra-operative, from intubation time to extubation time
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- ModerateNMB: This group underwent moderate neuromuscular blockade, defined as 1-2 twitches, in the beginning portion of the surgery or during the second portion of the surgery
Arm/Group | Deep NMB | ModerateNMB
Number analyzed (Participants) | 53 | 53
units on a scale | 5 [5 to 5] | 5 [5 to 5]
Statistical Analysis 1: Comparison: Deep NMB vs ModerateNMB; Test type: Superiority; p = 0.63, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Intraoperative (intubation time to extubation time)
Groups:
- Deep NMB: This group will underwent neuromuscular blockade, defined as post tetanic count (PTC) of 1 to 2, in the beginning portion or during the second portion of the surgery
Arm/Group | Deep NMB | Moderate NMB
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/53
Other Adverse Events (participants affected / at risk) | 0/53 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/86/NCT02812186/Prot_SAP_000.pdf